CLINICAL TRIAL: NCT03205982
Title: The Wise App Trial for Improving Health Outcomes in People Living With HIV
Brief Title: The Wise App Trial for Improving Health Outcomes in PLWH
Acronym: WiseApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Principal Investigator, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAQ9957; R01HS025071 (AHRQ)
Record Dates: First submitted 2017-05-24; First posted 2017-07-02 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: HIV/AIDS
Keywords: Wisepill; ART; PLWH
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): WiseApp that delivers fitness reminders
  Interventions: Behavioral: Wise app with fitness reminders
- Intervention (Experimental): WiseApp that delivers medication adherence reminders
  Interventions: Behavioral: Wise app with medication adherence reminders

INTERVENTIONS:
Behavioral: Wise app with medication adherence reminders — The Intervention group will receive the Wise app that delivers medication adherence reminders.
  Arms: Intervention
Behavioral: Wise app with fitness reminders — The control group will receive the Wise app with fitness reminders
  Arms: Control

SUMMARY:
The overall goal of this study is to design a user-centered design app linked to a smart pill box for people living with HIV (PLWH) and evaluate its effects in a randomized controlled trial. The proposed trial is scientifically significant in representing a principled and systematic effort to test the efficacy of a smartphone intervention linked to a smart pill box for antiretroviral (ART) adherence in PLWH in the United States (US). Guided by a strong theoretical framework building on earlier user-centered design work and integrating a real-time monitoring device, this work has the potential to improve ART adherence in PLWH and have a sustainable public health impact.

DETAILED DESCRIPTION:
Human Immunodeficiency virus (HIV) continues to affect 1.2 million Americans. Achieving viral suppression through adherence to antiretroviral (ART) therapy is a critical determinant of successful transmission prevention and long-term outcomes in HIV-infected patients. However only about 25% of persons living with HIV (PLWH) in the US are virally suppressed, demonstrating the need for effective interventions that enhance ART adherence. mHealth is a tool that has proven useful in supporting behavior change, but most mHealth tools for PLWH have not been well-developed or evaluated. Given the dearth of useful and likeable apps, the need for improving medication adherence in PLWH, and the great promise of mHealth, the investigators propose to build and test a user-centered smartphone app linked to a smart pill box targeting ART adherence in PLWH. Self-report of medication adherence is often criticized since it typically overestimated adherence especially in unmasked trials. Current adherence assessments, such as patient recall, pill counts and pharmacy refill data, typically detect missed doses long after they occur. This study will use real-time, wireless monitoring strategies via the Wisepill dispenser, for measuring ART adherence.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HIV
* Report past 30 days adherence of 80% or less as measured using the Visual Analogue Scale (VAS), or have a viral load of over 400 copies/mL
* Be able to communicate and read in English or Spanish
* Live in the US
* Have a smartphone
* Be taking ART medications

Exclusion Criteria:

* Participation in any other mobile app study for PLWH, including text messaging studies
* Diagnosis of a clinical problem that would preclude someone from using a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, RN, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarez G, Sanabria G, Jia H, Cho H, Reynolds NR, Gradilla M, Olender S, Mohr DC, Schnall R. Do Walk Step Reminders Improve Physical Activity in Persons Living With HIV in New York City?-Results From a Randomized Clinical Trial. J Assoc Nurses AIDS Care. 2023 Nov-Dec 01;34(6):527-537. doi: 10.1097/JNC.0000000000000427. Epub 2023 Sep 25. PMID 37747318
- [Derived] Sanabria G, Bushover B, Ashrafnia S, Cordoba E, Schnall R. Understanding Physical Activity Determinants in an HIV Self-Management Intervention: Qualitative Analysis Guided by the Theory of Planned Behavior. JMIR Form Res. 2023 Sep 14;7:e47666. doi: 10.2196/47666. PMID 37707942
- [Derived] Flynn G, Jia H, Reynolds NR, Mohr DC, Schnall R. Protocol of the randomized control trial: the WiseApp trial for improving health outcomes in PLWH (WiseApp). BMC Public Health. 2020 Nov 25;20(1):1775. doi: 10.1186/s12889-020-09688-0. PMID 33238931
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 101 | 99
Completed | 77 | 76
Not Completed | 24 | 23
Not completed — Lost to Follow-up | 20 | 19
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Withdrawal by PI | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only 198 out of 200 participants were included in the analysis. Valid data was not collected for 2 intervention group participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 101 | 97 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is in years
  years | 49.34 (10.2) | 49.19 (10.9) | 49.26 (10.5)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants' reported gender identity regardless of sex at birth
  Participants
    Male | 67 | 39 | 106
    Female | 28 | 55 | 83
    Transgender Male | 2 | 0 | 2
    Transgender Female | 4 | 2 | 6
    Other (Unspecified) | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 24 | 51
  Not Hispanic or Latino | 74 | 73 | 147
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 71 | 75 | 146
  White | 8 | 5 | 13
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 17 | 12 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101 | 97 | 198
Antiretroviral (ART) Adherence Visual Analog Scale [Mean (Standard Deviation); unit: units on a scale] — This visual analog scale asked participants to indicate percentage of ART medications taken in the past 30 days on a scale ranging from 0 to 100 with higher values indicating more adherence. One participant in control group did not provide baseline data for this measure. Population: One participant in control group did not provide baseline data for this measure.
  units on a scale
    number analyzed (Participants) | 100 | 97 | 197
    (all) | 71.76 (26.14) | 66.84 (26.63) | 69.37 (26.43)

OUTCOME MEASURES:

1. Primary Outcome: Change in ART Adherence - Clever Cap
Description: The CleverCapTM dispenser will automatically record each time a participant opens the dispenser. We will collect adherence data each day from the start to the end of trial (day 1 to 6 months), and it is a count response (number of times taking medication each day).
Time Frame: Up to 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Times taking medication/day
Arm/Group | Control | Intervention
Number analyzed (Participants) | 101 | 97
Times taking medication/day | 0.385 (0.487) | 0.445 (0.497)
Statistical Analysis 1: Comparison: Control vs Intervention; Compares difference in adherence changes between Intervention and Control arms; Test type: Equivalence — If the difference (between treatment and control arm) is greater than the minimal clinically important difference (MCID), we consider the treatment arm is different from the control arm. MCID is calculated as 0.25-0.5* standard deviation (SD). Conversely, the equivalence margin is the biggest difference (between 2 arms) to be considered no difference between 2 arms. Therefore, the equivalence margin should be smaller than MCID, i.e., it should be smaller than the smallest possible MCID; p < 0.0001, Mixed Models Analysis; generalized linear mixed model with logit link (logistic model); Odds Ratio (OR) = 0.9943, 95% CI 2-sided [0.993 to 0.995], Standard Error of Mean 0.0005

2. Secondary Outcome: Change in Score on the Center for Adherence Support Evaluation (CASE) Index
Description: The CASE Adherence Index is an easy to administer instrument that provides an alternative method for assessing ART adherence in clinical settings. Items are scored such that higher values indicate better adherence, minimum score is 3 and the maximum total score is 16. Scores of 11 or higher on this index indicate good adherence (Cronbach's α= 0.79).
Time Frame: Baseline, 3 month follow up, and 6 month follow up
Population: Only 198 out of 200 participants were included in the analysis. Valid data was not collected for 2 intervention group participants. In addition, the number of participants analyzed at each timepoint and for each group varied due to study attrition; participants missed visits, were lost to follow-up, and there were corona virus disease (COVID-19) restrictions in place.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 101 | 97
score on a scale
  Baseline | 9.099 (3.129) | 8.557 (2.926)
  3-Month Follow-up: number analyzed (Participants) | 84 | 81
  3-Month Follow-up | 10.667 (3.458) | 10.099 (3.345)
  6-Month Follow-up: number analyzed (Participants) | 77 | 76
  6-Month Follow-up | 10.714 (3.268) | 10.197 (3.533)

3. Secondary Outcome: Change in Cluster of Differentiation 4 (CD4) Count
Description: Using blood samples obtained during study visits, CD4 count will be used to asses ART adherence
Time Frame: Baseline, 3 month follow up, and 6 month follow up
Population: The number of participants analyzed at each timepoint and for each group varied due to study attrition; participants missed visits, were lost to follow-up, and there were COVID-19 restrictions in place.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Control | Intervention
Number analyzed (Participants) | 84 | 89
cells/mm^3
  Baseline | 5.972 (1.102) | 6.060 (0.806)
  3-Month Follow-up: number analyzed (Participants) | 83 | 80
  3-Month Follow-up | 5.811 (1.389) | 6.102 (0.838)
  6-Month Follow-up: number analyzed (Participants) | 76 | 76
  6-Month Follow-up | 5.772 (1.341) | 5.974 (0.941)

4. Secondary Outcome: Change in Viral Load
Description: Using blood samples obtained during study visits, viral load levels will be used to asses ART adherence.
Time Frame: Baseline, 3 month follow up, and 6 month follow up
Population: Only 198 out of 200 participants were included in the analysis. Valid data was not collected for 2 intervention group participants. In addition, the number of participants analyzed at each timepoint and for each group varied due to study attrition; participants missed visits, were lost to follow-up, and there were COVID-19 restrictions in place.
Measure: Mean (Standard Deviation); unit: copies/ml
Arm/Group | Control | Intervention
Number analyzed (Participants) | 101 | 97
copies/ml
  Baseline | 0.634 (0.484) | 0.567 (0.498)
  3-Month Follow-up: number analyzed (Participants) | 84 | 81
  3-Month Follow-up | 0.536 (0.502) | 0.444 (0.5)
  6-Month Follow-up: number analyzed (Participants) | 77 | 76
  6-Month Follow-up | 0.558 (0.5) | 0.5 (0.503)

5. Secondary Outcome: Change in Number of Primary Care Visits
Description: This will be measured by the self-reported number of primary care visits.
Time Frame: Baseline, 3 months, and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: primary care appointments
Arm/Group | Control | Intervention
Number analyzed (Participants) | 98 | 95
primary care appointments
  Baseline | 1.153 (0.484) | 1.084 (0.315)
  3-Month Follow-up: number analyzed (Participants) | 82 | 81
  3-Month Follow-up | 1.207 (0.561) | 1.111 (0.316)
  6-Month Follow-up: number analyzed (Participants) | 77 | 75
  6-Month Follow-up | 1.208 (0.592) | 1.24 (0.612)

6. Secondary Outcome: Change in Score on the Engagement With Health Care Provider Scale
Description: The Engagement with Health Care Provider 13-item Scale will be administered over the course of the trial to evaluate how participants' engagement with their health care providers changes their health care access overall. Items are scored such that higher scores indicate a more negative relationship with their health care provider. The minimum total score is 13 and the maximum total score is 52.
Time Frame: Baseline, 3 months, and 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 101 | 97
score on a scale
  Baseline | 17.386 (8.158) | 18.186 (8.121)
  3-Month Follow-up: number analyzed (Participants) | 84 | 81
  3-Month Follow-up | 16.607 (6.429) | 18.038 (8.528)
  6-Month Follow-up: number analyzed (Participants) | 77 | 76
  6-Month Follow-up | 18.221 (7.918) | 18.039 (8.589)

7. Secondary Outcome: Change in Score on the Perceived Ease of Use and Potential Usefulness Questionnaire
Description: Technology Acceptance: Perceived Ease of Use and Potential Usefulness 14-item Questionnaire provides a method for assessing participants' perception of the usefulness of the technology. Items are scored such that higher values indicate more positive perception. The minimum total score is 0 and the maximum total score is 70.
Time Frame: Baseline, 3 month follow up and 6 month follow up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 101 | 97
score on a scale
  Baseline | 2.053 (0.871) | 2.044 (0.950)
  3-Month Follow-up: number analyzed (Participants) | 84 | 81
  3-Month Follow-up | 1.807 (0.734) | 1.762 (0.826)
  6-Month Follow-up: number analyzed (Participants) | 77 | 76
  6-Month Follow-up | 1.861 (0.959) | 1.692 (0.733)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Description: All 200 participants were included in the adverse events analysis.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT03205982/Prot_SAP_000.pdf